CLINICAL TRIAL: NCT02541604
Title: An Early-Phase, Multicenter, Open-Label Study of the Safety and Pharmacokinetics of Atezolizumab (MPDL3280A) In Pediatric and Young Adult Patients With Previously Treated Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Preliminary Efficacy of Atezolizumab (Anti-Programmed Death-Ligand 1 [PD-L1] Antibody) in Pediatric and Young Adult Participants With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate because limited investigational agent activity was observed.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29664; 2014-004697-41 (EudraCT Number)
Record Dates: First submitted 2015-08-18; First posted 2015-09-04 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Atezolizumab (Experimental): Participants received intravenous (IV) infusion of atezolizumab (maximum 1200 milligrams [mg]) on Day 1 of each 21-day cycle.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab was administered as IV infusion (maximum 1200 mg) on Day 1 of each 21-day cycle.
  Other Names: RO5541267; MPDL3280A; Tecentriq

SUMMARY:
This early phase, multicenter, open-label, single-arm study evaluated the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary efficacy of atezolizumab in pediatric and young adult participants with solid tumors for which prior treatment was proven to be ineffective.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric solid tumor (including Hodgkin's and Non-Hodgkin's lymphoma), for which prior treatment had proven to be ineffective (that is, relapsed or refractory) or intolerable
* Disease that is measurable as defined by RECIST v1.1, mINRC, Revised Response Criteria for Malignant Lymphoma, RANO criteria (as appropriate) or evaluable by nuclear medicine techniques, immunocytochemistry techniques, tumor markers, or other reliable measures
* Archival tumor tissue block or 15 freshly cut, unstained, serial slides available for submission, or willingness to undergo a core or excisional biopsy prior to enrollment (fine-needle aspiration, brush biopsy, and lavage samples are not acceptable).

Participants with fewer than 15 slides available may be eligible for study entry following discussion with Medical Monitor

* Lansky Performance Status (participants less than [<] 16 years old) or Karnofsky Performance Status (participants greater than or equal to [>=] 16 years old) >=50
* Life expectancy >=3 months, in the investigator's judgment
* Adequate hematologic and end organ function, confirmed by laboratory results obtained within 28 days prior to initiation of study drug

Exclusion Criteria:

* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases, except ATRT
* Treatment with high-dose chemotherapy and hematopoietic stem-cell rescue within 3 months prior to initiation of study drug
* Prior allogeneic hematopoietic stem-cell transplantation or prior solid-organ transplantation
* Treatment with chemotherapy (other than high-dose chemotherapy as described above) or differentiation therapy (such as retinoic acid) or immunotherapy (such as anti-GD2 antibody treatment) within 3 weeks prior to initiation of study drug or, if treatment included nitrosoureas, within 6 weeks prior to initiation of study drug
* Treatment with thoracic or mediastinal radiotherapy within 3 weeks prior to initiation of study drug
* Treatment with hormonal therapy (except hormone replacement therapy or oral contraceptives) or biologic therapy within 4 weeks or 5 half-lives, whichever is shorter, prior to initiation of study drug. This requirement may be waived at the investigator's request if the participant has recovered from therapeutic toxicity to the degree specified in the protocol, with approval of the Medical Monitor
* Treatment with a long-acting hematopoietic growth factor within 2 weeks prior to initiation of study drug or a short-acting hematopoietic growth factor within 1 week prior to initiation of study drug
* Treatment with investigational therapy (with the exception of cancer therapies as described above) within 4 weeks prior to initiation of study drug
* Treatment with a live vaccine or a live, attenuated vaccine (e.g., nasal spray of live attenuated influenza vaccine or FluMist®) within 4 weeks prior to initiation of study drug or anticipation that such treatment will be required during the study or within 5 months after the final dose of study drug
* Treatment with herbal cancer therapy within 1 week prior to initiation of study drug
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA4), anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin 2 [IL-2]) within 6 weeks or five drug elimination half-lives prior to Day 1 of Cycle 1, whichever is longer
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) at the time of initiation of study drug, or anticipated requirement for systemic immunosuppressive medications during the study
* Current treatment with therapeutic anticoagulants
* Any non-hematologic toxicity (excluding alopecia) from prior treatment that has not resolved to Grade less than or equal to (<=) 1 (per National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.0) at screening
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (30):
- United States (7):
  - Arkansas Children'S Hospital, Little Rock, Arkansas
  - Stanford University/Lucile Packard Children's Hospital, Palo Alto, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
- Alberta Children'S Hospital, Calgary, Alberta, Canada
- Rigshospitalet; BØRNEUNGEKLINIKKEN, Ambulatoriet for kræft- og Blodsygdomme hos børn og unge, København Ø, Denmark
- France (3):
  - Centre Léon Bérard, Institut d'Hémato-Oncologie Pédiatrique, Lyon
  - Institut Curie, Oncologie Pédiatrique, Paris
  - Institut Gustave Roussy; Service Pediatrique, Villejuif
- Klinik Johann Wolfgang von Goethe Uni, Frankfurt, Germany
- Schneider Children's Medical Center, Petah Tikva, Israel
- Italy (5):
  - Ospedale Pediatrico Bambino Gesù - IRCCS; Dipartimento di Onco-Ematologia Pediatrica, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini; Unità Operativa Oncologica Pediatrica, Genoa, Liguria
  - Fondazione IRCCS Istituto Nazionale dei Tumori; Struttura Complessa di Pediatria Oncologica, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliera di Padova; Clinica di Onco-ematologia pediatrica, Padua, Veneto
- Erasmus MC / location Sophia Kinderziekenhuis, Rotterdam, Netherlands
- Spain (4):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universitäts-Kinderspital; Abteilung für Onkologie, Zurich, Switzerland
- United Kingdom (5):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital For Children, Bristol
  - Leeds General Infirmary; Paediatric Oncology & Haematology, Leeds
  - The Royal Victoria Infirmary; Paediatric and Adolescent Oncology Unit, Newcastle upon Tyne
  - Royal Marsden Hospital; Pediatric Unit, Surrey

REFERENCES:
- [Derived] Nabbi A, Danesh A, Espin-Garcia O, Pedersen S, Wellum J, Fu LH, Paulson JN, Geoerger B, Marshall LV, Trippett T, Rossato G, Pugh TJ, Hutchinson KE. Multimodal immunogenomic biomarker analysis of tumors from pediatric patients enrolled to a phase 1-2 study of single-agent atezolizumab. Nat Cancer. 2023 Apr;4(4):502-515. doi: 10.1038/s43018-023-00534-x. Epub 2023 Apr 10. PMID 37038005
- [Derived] Geoerger B, Zwaan CM, Marshall LV, Michon J, Bourdeaut F, Casanova M, Corradini N, Rossato G, Farid-Kapadia M, Shemesh CS, Hutchinson KE, Donaldson F, Liao M, Caron H, Trippett T. Atezolizumab for children and young adults with previously treated solid tumours, non-Hodgkin lymphoma, and Hodgkin lymphoma (iMATRIX): a multicentre phase 1-2 study. Lancet Oncol. 2020 Jan;21(1):134-144. doi: 10.1016/S1470-2045(19)30693-X. Epub 2019 Nov 25. PMID 31780255
- [Derived] Shemesh CS, Chanu P, Jamsen K, Wada R, Rossato G, Donaldson F, Garg A, Winter H, Ruppel J, Wang X, Bruno R, Jin J, Girish S. Population pharmacokinetics, exposure-safety, and immunogenicity of atezolizumab in pediatric and young adult patients with cancer. J Immunother Cancer. 2019 Nov 21;7(1):314. doi: 10.1186/s40425-019-0791-x. PMID 31753029

RESULTS

PARTICIPANT FLOW:
Groups:
- COHORT 1: EWING SARCOMA
- COHORT 2: HODGKIN LYMPHOMA
- COHORT 3: NEUROBLASTOMA
- COHORT 4: NON HODGKIN LYMPHOMA
- COHORT 5: NON-RHABDOMYOSARCOMA SOFT TISSUE SARCOMA;
- COHORT 6: OSTEOSARCOMA
- COHORT 7: RHABDOMYOSARCOMA
- COHORT 8: WILMS TUMOR
- COHORT 9: OTHER TUMOR TYPES WITH DOCUMENTED PD-L1 EXPRESSION
- COHORT 10: OTHER TUMOR TYPES WITHOUT DOCUMENTED PD-L1 EXPRESSION
- COHORT 11: RHABDOID TUMOR
- COHORT 12: ATYPICAL TERATOID RHABDOID TUMOR
Period: Overall Study
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | COHORT 5 | COHORT 6 | COHORT 7 | COHORT 8 | COHORT 9 | COHORT 10 | COHORT 11 | COHORT 12
Started | 11 | 9 | 11 | 3 | 10 | 10 | 10 | 10 | 4 | 4 | 2 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 11 | 9 | 11 | 3 | 10 | 10 | 10 | 10 | 4 | 4 | 2 | 3
Not completed — Death | 6 | 5 | 7 | 2 | 9 | 8 | 9 | 9 | 3 | 4 | 2 | 3
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Medical condition may jeopardize safety | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | COHORT 5 | COHORT 6 | COHORT 7 | COHORT 8 | COHORT 9 | COHORT 10 | COHORT 11 | COHORT 12 | Total
Number analyzed (Participants) | 11 | 9 | 11 | 3 | 10 | 10 | 10 | 10 | 4 | 4 | 2 | 3 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.6 (3.3) | 14.2 (3.0) | 12.8 (9.4) | 19.0 (6.6) | 14.5 (6.5) | 17.1 (4.1) | 13.0 (8.5) | 12.6 (6.8) | 14.8 (1.0) | 11.3 (0.5) | 0.5 (0.7) | 7.3 (4.6) | 13.5 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 4 | 0 | 5 | 4 | 4 | 6 | 0 | 4 | 1 | 1 | 40
  Male | 6 | 3 | 7 | 3 | 5 | 6 | 6 | 4 | 4 | 0 | 1 | 2 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 2 | 0 | 0 | 1 | 16
  Not Hispanic or Latino | 7 | 5 | 7 | 2 | 5 | 6 | 6 | 6 | 2 | 3 | 2 | 0 | 51
  Unknown or Not Reported | 2 | 3 | 2 | 0 | 4 | 2 | 1 | 3 | 0 | 1 | 0 | 2 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 6
  White | 8 | 5 | 5 | 2 | 6 | 6 | 8 | 5 | 1 | 2 | 2 | 0 | 50
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 4 | 4 | 0 | 4 | 2 | 2 | 4 | 1 | 1 | 0 | 2 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response (Complete Response [CR] or Partial Response [PR]) as Determined by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Participants With Solid Tumors
Description: Note: In Cohort 5, the response was observed in a rhabdoid tumor. Participant was erroneously enrolled in the Non-rhabdomyosarcoma soft tissue sarcoma cohort.
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 1: Participants with ewing sarcoma
- Cohort 5: Participants with non-rhabdomyosarcoma soft tissue sarcoma
- Cohort 6: Participants with osteosarcoma.
- Cohort 7: Participants with rhabdomyosarcoma
- Cohort 8: Participants with wilms tumor
- Cohort 9: Participants with other tumor types with documented PD-L1 expression.
- Cohort 10: Participants with other tumor types without documented PD-L1 expression.
- Cohort 11: Participants with rhabdoid tumor.
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 4 | 4 | 2
Percentage | 0 | 10.0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using Modified International Neuroblastoma Response Criteria (mINRC) in Participants With Neuroblastoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 3: Participants with neuroblastoma.
Arm/Group | Cohort 3
Number analyzed (Participants) | 11
Percentage | 0

3. Primary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using Revised Response Criteria for Malignant Lymphoma for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 2: Participants with Hodgkin's lymphoma
- Cohort 4: Participants with non-Hodgkin's lymphoma
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 9 | 3
Percentage | 22.2 | 33.3

4. Primary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using Response Assessment in Neuro-Oncology (RANO) Criteria in Participants With Atypical Teratoid Rhabdoid Tumor (ATRT)
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 12: Participants with atypical teratoid rhabdoid tumor.
Arm/Group | Cohort 12
Number analyzed (Participants) | 3
Percentage | 0

5. Primary Outcome: Percentage of Participants With Clinical Benefit as Determined by the Investigator According to RECIST v1.1 Criteria in Participants With Osteosarcoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population (defined as patients who received any amount of study drug), in the Osteosarcoma cohort as per protocol. (Objective response for the other cohorts are measured with different response criteria, and these are described in Outcome Measures 1, 2, 3, and 4).
Measure: Number; unit: Percentage
Arm/Group | Cohort 6
Number analyzed (Participants) | 10
Percentage | 0

6. Primary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator Using RECIST v1.1 in Participants With Solid Tumors
Time Frame: Baseline until first documented occurrence of progressive disease, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 10: Participant with other tumor types without documented PD-L1 expression.
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 4 | 4 | 2
Months | 1.2 [0.6 to 1.4] | 1.3 [1.1 to 1.4] | 1.2 [0.7 to 1.8] | 1.1 [0.8 to 1.3] | 1.3 [1.1 to 1.5] | 1.2 [0.7 to 1.3] | 1.2 [1.1 to 10.1] | 0.7 [0.3 to 1.1]

7. Primary Outcome: PFS as Determined by the Investigator Using mINRC in Participants With Neuroblastoma
Time Frame: as for outcome 6
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 3
Number analyzed (Participants) | 11
Months | 2.6 [1.2 to 4.7]

8. Primary Outcome: PFS as Determined by the Investigator Using Revised Response Criteria for Malignant Lymphoma for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: as for outcome 6
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 9 | 3
Months | 2.8 [2.6 to 4.4] | 1.4 [1.1 to NA] — More than 50% patient was censored.

9. Primary Outcome: PFS as Determined by the Investigator Using RANO Criteria in Participants With ATRT
Time Frame: as for outcome 6
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 12
Number analyzed (Participants) | 3
Months | 1.4 [1.4 to 1.7]

10. Primary Outcome: Percentage of Participants Adverse Events, Serious Adverse Events and Adverse Events of Special Interest
Time Frame: From baseline up to approximately 42 months
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Arm/Group | Atezolizumab
Number analyzed (Participants) | 87
Percentage
  Adverse Events | 97.7
  Serious Adverse Events | 37.9
  Adverse Events of Special Interest | 44.8

11. Primary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab
Time Frame: Predose (PRD; 0 hours [hr]), 0.5 hr post-infusion (P-I; infusion duration=30-60 minutes) on Day (D) 1 of Cycle (Cy) 1 and 4 (1 Cy=21 days)
Population: Included PK population, defined as patients who had received any amount of study drug and had at least one serum concentration result available at clinical data cutoff. In the "<2 Age (Years)" Arm/Group, 1 participant died after study entry with 1 cycle, and the other participant died after two cycles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- <2 Age (Years): Participants <2 Age (Years)
- 2 to <12 Age (Years): Participants 2 to <12 Age (Years)
- 12 to <18 Age (Years): Participants 12 to <18 Age (Years)
- >=18 Age (Years): Participants >=18 Age (Years)
Arm/Group | <2 Age (Years) | 2 to <12 Age (Years) | 12 to <18 Age (Years) | >=18 Age (Years)
Number analyzed (Participants) | 2 | 26 | 34 | 18
ug/mL
  Cycle 1 | 105 (6.90) | 312 (28.7) | 337 (26.8) | 424 (26.9)
  Cycle 4: number analyzed (Participants) | 0 | 11 | 16 | 6
  Cycle 4 |  | 382 (16.4) | 373 (78.9) | 626 (29.2)

12. Primary Outcome: Minimum Serum Concentration (Cmin) of Atezolizumab
Time Frame: PRD (0 hr) on D1 of Cy2,3,4,8, 12, 16 (1 Cy=21 days) and every 8 cycles thereafter; at any time during visit at study drug discontinuation visit, at least 90 days (maximum 150 days) after the last dose of study drug (up to approximately 42 months)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | <2 Age (Years) | 2 to <12 Age (Years) | 12 to <18 Age (Years) | >=18 Age (Years)
Number analyzed (Participants) | 1 | 25 | 32 | 16
ug/mL
  Cycle 2 | 24.1 (NA) — Later cycles are NA because 1 participant died after study entry with 1 cycle, and the other participant died after two cycles. | 59.3 (31.4) | 56.5 (50.4) | 79.9 (52.7)
  Cycle 3: number analyzed (Participants) | 0 | 13 | 19 | 8
  Cycle 3 |  | 58.9 (234.4) | 85.0 (47.4) | 148 (48.9)
  Cycle 4: number analyzed (Participants) | 0 | 11 | 16 | 6
  Cycle 4 |  | 99.2 (36.4) | 113 (41.1) | 121 (80.4)
  Cycle 8: number analyzed (Participants) | 0 | 4 | 4 | 2
  Cycle 8 |  | 166 (19.8) | 145 (21.9) | 209 (8.10)

13. Primary Outcome: Atezolizumab Serum Concentration at Washout
Time Frame: At least 90 days (maximum 150 days) after last dose of study drug (up to approximately 42 months)
Population: Included PK population, defined as patients who had received any amount of study drug and had at least one serum concentration result available at clinical data cutoff.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Atezolizumab
Number analyzed (Participants) | 17
ug/mL | 1.91 (2815.1)

14. Primary Outcome: Area Under the Concentration-Time Curve (AUC) of Atezolizumab
Time Frame: PRD (0 hr), 0.5 hr P-I (infusion duration=30-60 minutes) on D1 of Cy1; at any time during visit on Cy1D8 (1 Cy=21 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ugxday/mL
Arm/Group | <2 Age (Years) | 2 to <12 Age (Years) | 12 to <18 Age (Years) | >=18 Age (Years)
Number analyzed (Participants) | 2 | 29 | 38 | 18
ugxday/mL | 1130 (5.28) | 2209 (21.3) | 2816 (17.7) | 3579 (28.4)

15. Primary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Time Frame: PRD (0 hr) on D1 of Cy1,2,3,4,8,12,16 (1 Cy=21 days) & every 8 cycles thereafter; at any time during visit on Cy1D8, study drug discontinuation, at least 90 days (maximum 150 days) after last dose of study drug (up to approximately 42 months)
Population: The baseline ADA-evaluable population included patients who had a baseline ADA result. The post-baseline ADA-evaluable population included patients who had at least one post-baseline ADA result and had received at least one dose of that study treatment. Patients never dosed and patients without valid ADA records were not included in the analysis.
Measure: Number; unit: Percentage
Arm/Group | Atezolizumab
Number analyzed (Participants) | 78
Percentage
  Baseline | 2.6
  Post-baseline: number analyzed (Participants) | 77
  Post-baseline | 14.3

16. Secondary Outcome: Duration of Response (DOR) as Determined by the Investigator Using RECIST v1.1 Criteria in Participants With Solid Tumors
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Months |  | 13.2 [NA to NA] — There was only 1 participant. |  |  |  |  |  |

17. Secondary Outcome: DOR as Determined by the Investigator Using mINRC in Participants With Neuroblastoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Arm/Group | Cohort 3
Number analyzed (Participants) | 0

18. Secondary Outcome: DOR as Determined by the Investigator Using Revised Response Criteria for Malignant Lymphoma for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Cohort 2: Participants with hodgkin lymphoma.
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 2 | 1
Months | NA [4.1 to NA] — Kaplan-Meier median estimate not reached. | NA [NA to NA] — Kaplan-Meier median estimate not reached.

19. Secondary Outcome: DOR as Determined by the Investigator Using RANO Criteria in Participants With ATRT
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug. No participants had an objective response in this cohort.
Arm/Group | Cohort 12
Number analyzed (Participants) | 0

20. Secondary Outcome: Overall Survival (OS)
Time Frame: Baseline until death (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab
Number analyzed (Participants) | 87
Months | 7.4 [5.3 to 9.6]

21. Secondary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using Immune-Modified RECIST v1.1 for Participants With Other Solid Tumors
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 5: Participants with non-rhabdomyosarcoma.
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 4 | 4 | 2 | 3
Percentage | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using Immune-Related Response Criteria (irRC) for Participants With Neuroblastoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Arm/Group | Cohort 3
Number analyzed (Participants) | 11
Percentage | 0

23. Secondary Outcome: Percentage of Participants With an Objective Response (CR or PR) as Determined by the Investigator Using irRC for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Number; unit: Percentage
Groups:
- Cohort 4: Participants with non-hodgkin lymphoma.
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 9 | 3
Percentage | 33.3 | 33.3

24. Secondary Outcome: PFS as Determined by the Investigator Using Immune-Modified RECIST v1.1 for Participants With Other Solid Tumors
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12
Number analyzed (Participants) | 11 | 10 | 10 | 10 | 10 | 4 | 4 | 2 | 3
Months | 1.3 [0.6 to 1.4] | 1.4 [1.3 to 3.7] | 1.2 [0.9 to 1.8] | 1.3 [1.1 to 1.8] | 1.4 [1.1 to 2.8] | 1.2 [0.7 to 1.3] | 1.2 [1.1 to 10.1] | 0.7 [0.3 to 1.1] | 6.9 [1.7 to 9.3]

25. Secondary Outcome: PFS as Determined by the Investigator Using irRC for Participants With Neuroblastoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 3
Number analyzed (Participants) | 11
Months | 6.9 [2.6 to 14.7]

26. Secondary Outcome: PFS as Determined by the Investigator Using irRC for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 9 | 3
Months | 6.5 [2.6 to NA] — More than 50% patient was censored. | 3.7 [1.4 to NA] — More than 50% patient was censored.

27. Secondary Outcome: DOR as Determined by the Investigator Using Immune-Modified RECIST v1.1 for Participants With Other Solid Tumors
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 5 | Cohort 6 | Cohort 7 | Cohort 8 | Cohort 9 | Cohort 10 | Cohort 11 | Cohort 12
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Months |  | 13.2 [NA to NA] — There was only 1 participant with response. |  |  |  |  |  |  |

28. Secondary Outcome: DOR as Determined by the Investigator Using irRC for Participants With Neuroblastoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug. No participants had response therefore no participants analyzed.
Arm/Group | Cohort 3
Number analyzed (Participants) | 0

29. Secondary Outcome: DOR as Determined by the Investigator Using irRC for Participants With Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma
Time Frame: Baseline until disease progression, or death from any cause, whichever occurs first (up to approximately 42 months)
Population: Included safety-evaluable population, defined as patients who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 2 | Cohort 4
Number analyzed (Participants) | 3 | 1
Months | NA [7.3 to NA] — Kaplan-Meier median estimate not reached. | NA [NA to NA] — Kaplan-Meier median estimate not reached.

30. Secondary Outcome: Optimal Dose of Atezolizumab in Pediatric Adult Participants
Description: Atezolizumab was administered on Day 1 only for a cycle duration of 3 weeks.
Time Frame: From baseline up to approximately 42 months
Measure: Number; unit: mg/kg
Groups:
- <18 Age (Years): Participants <18 Age (Years)
Arm/Group | <18 Age (Years)
Number analyzed (Participants) | 69
mg/kg | 15

31. Secondary Outcome: Optimal Dose of Atezolizumab in Young Adult Participants
Description: Atezolizumab was administered on Day 1 only for a cycle duration of 3 weeks.
Time Frame: From baseline up to approximately 42 months
Measure: Number; unit: mg
Arm/Group | >=18 Age (Years)
Number analyzed (Participants) | 18
mg | 1200

ADVERSE EVENTS:
Time Frame: From baseline up to approximately 42 months
Description: Adverse Events reporting is for the Safety Evaluable Population, defined as patients who received any amount of any component of study treatment.
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3 | COHORT 4 | COHORT 5 | COHORT 6 | COHORT 7 | COHORT 8 | COHORT 9 | COHORT 10 | COHORT 11 | COHORT 12
All-Cause Mortality (participants affected / at risk) | 6/11 | 5/9 | 7/11 | 2/3 | 9/10 | 8/10 | 9/10 | 9/10 | 3/4 | 4/4 | 2/2 | 3/3
Serious Adverse Events (participants affected / at risk) | 4/11 | 3/9 | 2/11 | 0/3 | 3/10 | 6/10 | 3/10 | 5/10 | 2/4 | 3/4 | 1/2 | 1/3
Other Adverse Events (participants affected / at risk) | 11/11 | 8/9 | 11/11 | 3/3 | 10/10 | 10/10 | 10/10 | 10/10 | 4/4 | 3/4 | 2/2 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=11) | COHORT 2 (N=9) | COHORT 3 (N=11) | COHORT 4 (N=3) | COHORT 5 (N=10) | COHORT 6 (N=10) | COHORT 7 (N=10) | COHORT 8 (N=10) | COHORT 9 (N=4) | COHORT 10 (N=4) | COHORT 11 (N=2) | COHORT 12 (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAPILLOEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCISION SITE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POSTOPERATIVE HYPOTENSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VITH NERVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUPERIOR VENA CAVA SYNDROME (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=11) | COHORT 2 (N=9) | COHORT 3 (N=11) | COHORT 4 (N=3) | COHORT 5 (N=10) | COHORT 6 (N=10) | COHORT 7 (N=10) | COHORT 8 (N=10) | COHORT 9 (N=4) | COHORT 10 (N=4) | COHORT 11 (N=2) | COHORT 12 (N=3)
ANAEMIA (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 3 (6) | 1 (1) | 5 (12) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FANCONI SYNDROME (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECZEMA EYELIDS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPSOCLONUS MYOCLONUS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHOTOPSIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (4) | 3 (3) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 3 (6) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 6 (7) | 2 (2) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (5) | 0 (0) | 4 (6) | 4 (5) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIP ULCERATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 1 (3) | 1 (2) | 0 (0) | 2 (2) | 4 (7) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
NONINFECTIVE GINGIVITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ODYNOPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL DISCHARGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (4) | 3 (6) | 2 (2) | 0 (0) | 3 (5) | 3 (4) | 1 (2) | 4 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AXILLARY PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER SITE ERYTHEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHILLS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 2 (3) | 2 (2) | 3 (3) | 0 (0) | 4 (13) | 6 (6) | 3 (3) | 6 (7) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
GENERALISED OEDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALAISE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 3 (5) | 3 (9) | 4 (5) | 2 (2) | 2 (5) | 8 (14) | 5 (6) | 4 (5) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
THIRST (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VACCINATION SITE OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA URETHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATOPHYTOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 4 (16) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VULVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL SWELLING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSTOMY COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 1 (3) | 3 (3) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AMYLASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANTITHROMBIN III DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (3) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CHLORIDE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CANDIDA TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CARDIAC MURMUR (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (6) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (3) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NOROVIRUS TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OXYGEN SATURATION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROTHROMBIN LEVEL DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VITAMIN K DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 2 (4) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (2) | 2 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR INFLAMMATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AMPUTATION STUMP PAIN (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (8) | 3 (3) | 1 (1) | 2 (3) | 2 (8) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHANTOM LIMB SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE BREAKAGE (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRUXISM (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
IRRITABILITY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLYCOSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OLIGURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (14) | 2 (2) | 1 (1) | 1 (1) | 5 (8) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IRREGULAR BREATHING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DISORDER OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PALMAR-PLANTAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORAL DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PITYRIASIS ROSEA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CENTRAL VENOUS CATHETERISATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EMBOLISM (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOUS THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PARAPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02541604/Prot_SAP_000.pdf